CLINICAL TRIAL: NCT05571436
Title: iCan Diabetes Self-Management and Prevention Support Group
Brief Title: iCan Diabetes Self-management and Prevention Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Seung-Yeon Lee, Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0532
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
Keywords: Diabetes Mellitus, Type 2; Prediabetes; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): iCan Diabetes Self-Management and Prevention Program
  Interventions: Behavioral: iCan Diabetes Self-management and Prevention Support Group

INTERVENTIONS:
Behavioral: iCan Diabetes Self-management and Prevention Support Group — Participants will be asked to attend six weekly sessions and complete pre-and post-assessments with an optional focus group.
  The intervention will cover the following topics: 1) Yes, iCan! - Affirmations and Empowerment, 2) The Language of Diabetes - Diabetes Synopsis, 3) Diabetes and Me - Management Strategies, 4) Extraordinary Health - Dream Team, 5) Food for Thought - Food Conscious, and 6) Discussion - Stories/Goals.
  Each session is composed of a Check-in, Affirmation/Empowerment Activity, Short Presentation, Q&A and Discussion, Goal setting, and Testing Healthy Snacks.

SUMMARY:
The purpose of this study is to test the feasibility and preliminary efficacy of the iCan Diabetes Self-Management and Prevention Support Group using a single arm clinical trial. The program is composed of six weekly sessions, and it will be implemented with 60 adults (aged 18 years or older) who have been diagnosed with type 2 diabetes or prediabetes and evaluated using mixed methods. A pre-test will be conducted before the program implementation and a post-test will be conducted three months after the pre-test. Focus groups will be conducted shortly after the last session to obtain feedback on the program. Between the last session and the post-test, weekly emails/texts will be sent to keep participants engaged and maximize retention rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or older
* Have been diagnosed with type 2 diabetes or prediabetes
* Can read, write, and speak in English

Exclusion Criteria:

* Attended a diabetes self-management program or diabetes prevention program within the last 3 months
* Plan to attend another diabetes self-management program or diabetes prevention program within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (A1C) | 3 months
  Glycemic control
Diabetes self-management behavior | 3 months
  Diabetes Self-Management Questionnaire (DSMQ) (16 items)

SECONDARY OUTCOMES:
Self-efficacy related to diabetes self-management | 3 months
  Diabetes Empowerment Scale (28 items)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yeon Lee, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No